CLINICAL TRIAL: NCT06398678
Title: Retrospective Evaluation of Anesthesia Management and Clinical Outcomes in Patients Undergoing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Anesthesia Management in Patients Undergoing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, ahmet kaya, assistant professor, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: MAIEAHANEST
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cytoreductive Surgery; Hyperthermic Intraperitoneal Chemotherapy; Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had undergone cytoreductive surgery.

SUMMARY:
A combined approach of cytoreductive surgery (SRC) and hyperthermic intraperitoneal chemotherapy (HIPEC) represents a potential treatment option for patients diagnosed with primary or secondary gastrointestinal or gynaecological malignancies with peritoneal involvement. While the surgical phase of the operation macroscopically addresses the cancerous tissue, the HIPEC phase targets the microscopic tumour cells that remain after surgery (1). The surgical procedure known as SRC and HIPEC is one of the most complex surgical procedures, presenting numerous challenges for both the surgical and anaesthesia teams. The haemodynamic, haematological and metabolic changes that occur before, during and in the early postoperative period are associated with an increased risk of morbidity and mortality. It is therefore crucial for anaesthesia management to maintain normovolemia during surgery, compensate for hypothermia in the surgical phase and hyperthermia in the HIPEC phase, and maintain metabolic and haemodynamic balance throughout the entire procedure.

The objective of this study was to retrospectively examine the anaesthesia management and clinical outcomes in patients who underwent cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC) in order to create literature information that can facilitate the early recognition and prevention of haemodynamic, haematological and metabolic problems that occur especially in the intraoperative and postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary or secondary gastrointestinal or gynecologic malignancies with peritoneal involvement.
* Over 18 years of age

Exclusion Criteria:

* Over 80 years of age
* those with heart, lung and liver diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include cases of patients over the age of 18 who underwent hyperthermic intraperitoneal chemotherapy with the closed method in accordance with the protocols determined by the Department of Surgical Oncology for 4 years retrospectively at the University of Health Sciences Şanlıurfa Mehmet Akif İnan Health Application and Research Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Anesthesia Management in Hyperthermic Intraperitoneal Chemotherapy | 01/01/2020 - 01/01/2024
  anaesthesia management in cytoreductive surgery and while hypertermic intraperitoneal chemotherapy
perioperative complications | during the operation
  The potential complications associated with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy will be identified from the documented records.
fluid transfusion amounts | during the operation
  The quantity of fluid transfusion administered to the patient during cytoreductive surgery and hyperthermic intraperitoneal chemotherapy will be determined from documented records in millilitres.
blood replacements | during the operation
  The quantity and type of blood and blood products transfused to the patient during cytoreductive surgery and hyperthermic intraperitoneal chemotherapy will be determined from documented records in millilitres.
procedure times | during the operation
  The duration of the surgical procedure applied to the patient during cytoreductive surgery and hyperthermic intraperitoneal chemotherapy will be determined from the documents recorded in minutes.
30-day mortality and morbidity | post-operative 30 days
  The morbidity and mortality rate observed in the patient within 30 days of cytoreductive surgery and hyperthermic intraperitoneal chemotherapy will be quantified as a percentage based on the documented records.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Turkey Sanliurfa Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaya A, Karahan MA. Retrospective evaluation of anesthesia management and clinical outcomes in patients undergoing cytoreductive surgery and hyperthermic intraperitoneal chemotherapy. BMC Anesthesiol. 2025 Jul 30;25(1):369. doi: 10.1186/s12871-025-03241-5. PMID 40739475